CLINICAL TRIAL: NCT00405938
Title: A Phase II Trial of Open-Label Bevacizumab Administered With Anastrozole or Fulvestrant as First-Line Therapy in Postmenopausal Hormone Receptor- Positive Metastatic Breast Cancer (With Trastuzumab in HER2-Positive Patients)
Brief Title: Bevacizumab Given With Either Anastrozole or Fulvestrant With Trastuzumab for Postmenopausal Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 86
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Breast cancer; Metastatic breast cancer; Bevacizumab; Anastrozole; Fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Anastrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab/anastrozole (Experimental): Bevacizumab 10mg/kg IV every 2 weeks [patients who are also receiving trastuzumab have the option to receive their bevacizumab at 15 mg/kg every 3 weeks instead of 10 mg/kg every 2 weeks (see Trastuzumab section below)] and anastrozole (1 mg orally daily). Treatment will be given in 4-week cycles.
  Interventions: Drug: Bevacizumab; Drug: Anastrozole
- Bevacizumab/fulvestrant (Experimental): Bevacizumab/fulvestrant (with trastuzumab in HER2+ patients). Bevacizumab 10mg/kg IV every 2 weeks [patients who are also receiving trastuzumab have the option to receive their bevacizumab at 15 mg/kg every 3 weeks instead of 10 mg/kg every 2 weeks (see Trastuzumab section below)] fulvestrant (500 mg IM on Day 1 of Cycle 1, followed by 250 mg IM of fulvestrant on Day 15 of Cycle 1. On Day 1 of Cycle 2 and the first day of all subsequent cycles thereafter, patients in this treatment arm will receive 250 mg IM of fulvestrant). Treatment will be given in 4-week cycles.
  Interventions: Drug: Bevacizumab; Drug: Fulvestrant

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 10mg/kg IV every 2 weeks
  Other Names: Avastin
Drug: Anastrozole — anastrozole (1 mg orally daily)
  Other Names: Arimidex
  Arms: Bevacizumab/anastrozole
Drug: Fulvestrant — fulvestrant (500 mg IM on Day 1 of Cycle 1, followed by 250 mg IM of fulvestrant on Day 15 of Cycle 1. On Day 1 of Cycle 2 and the first day of all subsequent cycles thereafter, patients in this treatment arm will receive 250 mg IM of fulvestrant).
  Other Names: Faslodex
  Arms: Bevacizumab/fulvestrant

SUMMARY:
This is a phase II trial combining bevacizumab with either fulvestrant or anastrozole with trastuzumab in the treatment of metastatic breast cancer in postmenopausal women. It is hoped that these combinations will keep the cancer from growing and spreading further.

DETAILED DESCRIPTION:
Regimen A: Bevacizumab/anastrozole (with trastuzumab in HER2+ patients). Bevacizumab 10mg/kg IV every 2 weeks [patients who are also receiving trastuzumab have the option to receive their bevacizumab at 15 mg/kg every 3 weeks instead of 10 mg/kg every 2 weeks (see Trastuzumab section below)] and anastrozole (1 mg orally daily). Treatment will be given in 4-week cycles. Response assessments will be performed after 2 cycles. Patients who respond to treatment or have stable disease will continue to be evaluated every 2 cycles. After 6 months, response assessment will occur every 3 months. A patient may remain on study if radiation is deemed necessary and appropriate, provided that there are other sites of measurable disease outside the field of radiation that may be followed. Treatment occurs until disease progression. Patients will be selected for this treatment arm per the following guidelines: >=12 months from adjuvant endocrine therapy OR >=12 months from adjuvant aromatase inhibitors OR Endocrine therapy naive OR Prior tamoxifen exposure or tamoxifen intolerance

Regimen B: Bevacizumab/fulvestrant (with trastuzumab in HER2+ patients). Bevacizumab 10mg/kg IV every 2 weeks [patients who are also receiving trastuzumab have the option to receive their bevacizumab at 15 mg/kg every 3 weeks instead of 10 mg/kg every 2 weeks (see Trastuzumab section below)] fulvestrant (500 mg intramuscular on Day 1 of Cycle 1, followed by 250 mg intramuscular of fulvestrant on Day 15 of Cycle 1. On Day 1 of Cycle 2 and the first day of all subsequent cycles thereafter, patients in this treatment arm will receive 250 mg intramuscularly of fulvestrant). Treatment will be given in 4-week cycles. Response assessments will be performed after 2 cycles. Patients who respond to treatment or have stable disease will continue to be evaluated every 2 cycles. After 6 months, response assessment will occur every 3 months. A patient may remain on study if radiation is deemed necessary and appropriate, provided that there are other sites of measurable disease outside the field of radiation that may be followed. Treatment occurs until disease progression. Patients will be selected for this treatment arm per the following guidelines: <12 months from adjuvant aromatase inhibitor therapy OR Intolerant of aromatase inhibitors OR Disease progression on adjuvant aromatase inhibitors OR Physician discretion

Trastuzumab: Patients in Treatment Arm A or Treatment Arm B who have FISH HER2+ or IHC3+ breast cancer will also receive treatment with trastuzumab in addition to their treatment with the combination of bevacizumab with either anastrozole or fulvestrant. Trastuzumab will be administered ONLY to patients with HER2+ breast cancer (FISH-positive or IHC3+). An 8 mg/kg loading dose of IV trastuzumab will be administered on Day 1, followed by doses of 6 mg/kg IV trastuzumab once every 3 weeks. These patients will have the option of receiving their bevacizumab doses at 15 mg/kg every 3 weeks rather than 10 mg/kg every 2 weeks (if they prefer to keep their bevacizumab dosing schedule consistent with their trastuzumab dosing schedule so that the number of visits they must make to the study site is minimized). The dosing schedules for anastrozole (for HER2+ patients in Treatment Arm A) and fulvestrant (for HER2+ patients in Treatment Arm B) will not change.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal breast cancer (adenocarcinoma) estrogen (ER)and/or progesterone (PR) receptor positive that is locally advanced or locally recurrent and not able to be surgically removed OR with measurable and/or disease that is able to be assessed including isolated bone metastasis
* Female patients 18 years or older
* Documentation of ER+ and/or PR+
* No prior chemotherapy or hormone therapy for metastatic breast cancer or inoperable breast cancer that is locally recurrent or locally advanced
* Measurable or evaluable disease
* Radiation therapy to painful bone lesions or impending fractures is allowed as long as there is measurable or evaluable disease outside the radiated area.
* Must have adequate bone marrow, renal and liver function
* Patients receiving prior treatment with an anthracycline based chemotherapy must have a normal left ventricle ejection fraction

Exclusion Criteria:

* No metastatic disease to the Central Nervous System
* No history of myocardial infarction (MI), stroke or transient ischemic attacks in the last 6 months
* No symptoms of peripheral vascular disease
* No history of abdominal fistula, gastrointestinal perforation or intrabdominal abscess in the past 6 months
* No known hypersensitivity to phosphate, trehalose or polysorbate
* No serious non-healing wound, ulcer or bone fracture
* No uncontrolled high blood pressure or history of hypertensive crisis
* No New York Hear Association class II congestive heart failure
* No extensive cancer involvement of the liver or lungs
* No history of significant psychiatric disorders
* No significant vascular disease

There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-11; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (11):
- United States (11):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Sletten Cancer Institute, Great Falls, Montana
  - Chattanooga Oncology & Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Background] Yardley DA, Burris HA 3rd, Clark BL, Shipley D, Rubin M, Barton J Jr, Arrowsmith E, Hainsworth JD. Hormonal therapy plus bevacizumab in postmenopausal patients who have hormone receptor-positive metastatic breast cancer: a phase II Trial of the Sarah Cannon Oncology Research Consortium. Clin Breast Cancer. 2011 Jun;11(3):146-52. doi: 10.1016/j.clbc.2011.03.010. Epub 2011 Apr 20. PMID 21665134

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab/Fulvestrant: Bevacizumab/fulvestrant (with trastuzumab in HER2+ patients). Bevacizumab 10mg/kg IV every 2 weeks [patients who are also receiving trastuzumab have the option to receive their bevacizumab at 15 mg/kg every 3 weeks instead of 10 mg/kg every 2 weeks (see Trastuzumab section below)] fulvestrant (500 mg intramuscular on Day 1 of Cycle 1, followed by 250 mg intramuscular of fulvestrant on Day 15 of Cycle 1. On Day 1 of Cycle 2 and the first day of all subsequent cycles thereafter, patients in this treatment arm will receive 250 mg intramuscular of fulvestrant). Treatment will be given in 4-week cycles.
Period: Overall Study
Arm/Group | Bevacizumab/Anastrozole | Bevacizumab/Fulvestrant
Started | 38 | 41
Completed | 38 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab/Anastrozole | Bevacizumab/Fulvestrant | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Continuous [Median (Full Range); unit: years] | 62 [37 to 85] | 63 [48 to 88] | 63 [37 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 79
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Description: Progression Free Survival (PFS) is defined as the interval, in months, from the date of first treatment to the date of disease progression or death, whichever occurred first.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Anastrozole | Bevacizumab/Fulvestrant
Number analyzed (Participants) | 38 | 41
months | 21 [14 to NA] — Upper limit not reached due to patients remaining on treatment at time of analysis. | 9 [5 to 13]

2. Secondary Outcome: Objective Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment (CR+PR). The response categories were assigned using RECIST criteria. Complete Response (CR) = Disappearance of all target lesions ; Partial Response (PR) = >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab/Anastrozole | Bevacizumab/Fulvestrant
Number analyzed (Participants) | 38 | 41
Participants | 18 | 11

ADVERSE EVENTS:
Arm/Group | Bevacizumab/Anastrozole | Bevacizumab/Fulvestrant
Serious Adverse Events (participants affected / at risk) | 10/38 | 12/41
Other Adverse Events (participants affected / at risk) | 38/38 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Anastrozole (N=38) | Bevacizumab/Fulvestrant (N=41)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
cTnI (Cardiac disorders) | 0 (0) | 1 (1) — Elevated cardiac enzymes
Superventricular Arrhythmia - Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Infection - Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Pain - Cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Mood Alteration - Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CNS Ischemia (Nervous system disorders) | 1 (1) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection - Wound (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - Abdomen (Surgical and medical procedures) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Weakness (General disorders) | 1 (1) | 0 (0)
Restrictive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Anastrozole (N=38) | Bevacizumab/Fulvestrant (N=41)
Anorexia (Gastrointestinal disorders) | 7 (23) | 7 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (121) | 10 (34)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
AST (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Bilirubin (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Cardiac Genral, Other (Decreased LVEF) (Cardiac disorders) | 2 (2) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (11) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 8 (29)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 3 (20)
Dehydration (Gastrointestinal disorders) | 2 (2) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 9 (18) | 9 (12)
Dizziness (Nervous system disorders) | 4 (9) | 9 (22)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 9 (13)
Edema - Limb (Blood and lymphatic system disorders) | 5 (46) | 7 (33)
Edema - NOS (Blood and lymphatic system disorders) | 3 (23) | 0 (0)
Fatigue (General disorders) | 22 (168) | 30 (170)
Fever (General disorders) | 4 (4) | 3 (5)
Pain - Head (General disorders) | 17 (53) | 3 (3)
Heartburn (Gastrointestinal disorders) | 4 (17) | 7 (27)
Hemoglobin (Blood and lymphatic system disorders) | 13 (57) | 12 (44)
Hemorrhage - Nose (Blood and lymphatic system disorders) | 8 (14) | 10 (21)
Hemorrhoids (Gastrointestinal disorders) | 2 (10) | 0 (0)
Hot Flashes (Endocrine disorders) | 13 (51) | 8 (23)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (8) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7) | 3 (7)
Hypertension (Cardiac disorders) | 18 (70) | 20 (110)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypotension (Cardiac disorders) | 0 (0) | 5 (6)
Infection - Dental (Infections and infestations) | 0 (0) | 3 (6)
Infection - Ear (Infections and infestations) | 2 (6) | 0 (0)
Infection - Sinus (Infections and infestations) | 4 (16) | 4 (5)
Infection - Skin (Infections and infestations) | 2 (2) | 0 (0)
Infection - Bladder (Infections and infestations) | 6 (9) | 3 (6)
Infection - Pulmonary (Infections and infestations) | 4 (5) | 0 (0)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Insomnia (General disorders) | 5 (13) | 4 (10)
Leukopenia (Blood and lymphatic system disorders) | 5 (13) | 8 (19)
Lymphedema (Blood and lymphatic system disorders) | 2 (7) | 0 (0)
Mood Alteration - Anxiety (Psychiatric disorders) | 5 (18) | 6 (18)
Mood Alteration - Depression (Psychiatric disorders) | 4 (19) | 4 (26)
Mood Alteration - NOS (Psychiatric disorders) | 3 (11) | 0 (0)
Mucositis/Stomatitis (Gastrointestinal disorders) | 4 (4) | 7 (20)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (9) | 5 (14)
Nausea (Gastrointestinal disorders) | 14 (48) | 12 (44)
Neuropathy - Motor (Nervous system disorders) | 2 (5) | 0 (0)
Neuropathy - Sensory (Nervous system disorders) | 7 (12) | 9 (15)
Neutrophils (Blood and lymphatic system disorders) | 2 (46) | 3 (4)
Pain - Abdomen (General disorders) | 4 (22) | 0 (0)
Pain - Back (General disorders) | 8 (39) | 12 (24)
Pain - Bladder (General disorders) | 2 (2) | 0 (0)
Pain - Bone (General disorders) | 4 (9) | 7 (61)
Pain - Breast (General disorders) | 2 (2) | 0 (0)
Pain - Chest Wall (General disorders) | 6 (6) | 5 (12)
Pain - Ear (General disorders) | 2 (6) | 0 (0)
Pain - Joint (General disorders) | 11 (37) | 10 (28)
Pain - Limb (General disorders) | 13 (81) | 12 (32)
Pain - Muscle (General disorders) | 4 (10) | 3 (9)
Pain - Neck (General disorders) | 3 (24) | 0 (0)
Pain - NOS (General disorders) | 2 (9) | 0 (0)
Pain - Pelvis (General disorders) | 0 (0) | 3 (10)
Platelets (Blood and lymphatic system disorders) | 8 (41) | 4 (11)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 13 (97) | 18 (91)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 4 (14) | 5 (6)
Renal Insufficiency (Renal and urinary disorders) | 2 (2) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 (32) | 7 (38)
Rigor/Chills (General disorders) | 2 (2) | 3 (8)
Taste Alteration (Gastrointestinal disorders) | 3 (20) | 0 (0)
Sweating (General disorders) | 0 (0) | 4 (11)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 (13) | 0 (0)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (28)
Vomiting (Gastrointestinal disorders) | 7 (14) | 5 (7)
Weakness (General disorders) | 5 (11) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 4 (32) | 3 (4)
Wound Complication (Surgical and medical procedures) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.